CLINICAL TRIAL: NCT03765320
Title: Impact of Peritoneal Closure and Retroperitoneal Drainage on Patients Who Underwent Laparotomic Retroperitoneal Lymph Node Dissection for Early Gynecological Cancer
Brief Title: Impact of Peritoneal Closure and Retroperitoneal Drainage on Patients Who Underwent Laparotomic Retroperitoneal Lymph Node Dissection
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 107150-E
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Lymphocele; Gynecologic Cancer
MeSH Terms: conditions — Lymphocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Peritoneal closure — Peritoneal closure after pelvic lymph node dissection for early gynecologic cancer
Procedure: Retroperitoneal drainage — Retroperitoneal drainage after pelvic lymph node dissection for early gynecologic cancer

SUMMARY:
To elucidate whether peritoneal closure and retroperitoneal drainage can benefit clinical outcome of early gynecologic cancer patients who underwent retroperitoneal lymph node dissection.

DETAILED DESCRIPTION:
To elucidate whether peritoneal closure and retroperitoneal drainage can benefit clinical outcome of early gynecologic cancer patients who underwent retroperitoneal lymph node dissection by reviewing the medical records of patients who underwent retroperitoneal lymph node dissection for stage I or II gynecological cancer in Far Eastern Memorial Hospital, January 2011~December 2017.

ELIGIBILITY:
Inclusion Criteria:

* Stage I or stage II gynecologic cancer (including cervical cancer, endometrial cancer, ovarian cancer, and fallopian tube cancer)
* Underwent laparotomic gynecologic oncologic surgery, including retroperitoneal lymphadenectomy.

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early gynecologic cancer patients who underwent retroperitoneal lymph node dissection in Far Eastern Memorial Hospital between January 2011 and December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Factors predicting lymphocele occurrence | 10 year
  To find independent factors that can predict lymphocele occurrence in patients who underwent laparotomic gynecologic oncologic surgery

SECONDARY OUTCOMES:
Factors predicting surgical complication | 10 years
  To find independent factors that can predict occurrence of surgical complication in patients who underwent laparotomic gynecologic oncologic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided